CLINICAL TRIAL: NCT05629130
Title: Embolization in Hereditary Coagulopathies
Acronym: EHCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63452822.1.0000.0068
Record Dates: First submitted 2022-09-28; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-09

CONDITIONS: Hemophilia; Embolization; Hemarthrosis; Clotting Factor Deficiency; Synovitis; Arthropathy
MeSH Terms: conditions — Hemophilia A; Hemarthrosis; Synovitis; Joint Diseases | interventions — Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: longitudinal, prospective study.
Masking Description: no masking - all treatement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization (Experimental): embolization procedure (superselective embolization of target arteries with spherical microparticles Embosphere 100-300 micrometers (Biosphere Medical, Roissy, France) of the affected joint, until partial vascular stasis and decharacterization of pathological synovial enhancement.
  Interventions: Device: embolization with spherical microparticles embosphere

INTERVENTIONS:
Device: embolization with spherical microparticles embosphere — embolization of affected joints with spherical microparticles embosphere

SUMMARY:
This is a longitudinal, prospective study, which will include 30 subjects with hereditary coagulopathies, with arthropathy, chronic synovitis resulting from hemarthrosis of the elbows, knees and/or ankles followed up at the Centro de Hemofilia HCFMUSP, after approval by the ethics and research committee.

They will undergo imaging tests (X-rays and Magnetic Resonance of knee, elbow, or ankle), physical, pain, quality of life and functional assessments (Hemophilia Joint Health Score, Functional Independence Score in Hemophilia, Perimeter, Test Timed up and Go, 30 second sit and stand test, Haemophilia - Adult - Quality of Life questionnaire (HAEM-A-QoL), Knee Injury and Osteoarthritis Outcome Score, EQ-5D, numerical rating scale for pain and embolization procedure (superselective embolization of target arteries with spherical microparticles Embosphere 100-300 micrometers (Biosphere Medical, Roissy, France), until partial vascular stasis and decharacterization of pathological synovial enhancement.

These evaluations will be performed at baseline, 1, 3, 6, 12, 24, 36, 48 and 60 months after the procedure.

DETAILED DESCRIPTION:
Longitudinal, prospective study, which will include 30 subjects with hereditary coagulopathies, with arthropathy, chronic synovitis resulting from hemarthrosis of the elbows, knees and/or ankles followed up at the Centro de Hemophilia do Hospital das Clinicas, Faculdade de Medicina da Universidade de São Paulo, i.e. HC-FMUSP), after approval by the ethics and research committee and registry at the clinical trials.

Patients will be evaluated by imaging (X-rays and Magnetic Resonance of the affected joint, i.e., knee, elbow, and/or ankle); physical and functional assessments (Hemophilia Joint Health Score, Functional Independence Score in Hemophilia, Perimeter of the affected joint(s), Test Timed up and Go, 30 second sit and stand test, Knee Injury and Osteoarthritis Outcome Score (KOOS); quality of life (Haemophilia - adult - quality of life questionnaires (HAEM-A-QoL), Knee Injury and Osteoarthritis Outcome Score (KOOS), EQ-5D; pain measured by numerical rating scale.

Volunteers will be submitted to embolization procedure (superselective embolization of target arteries with spherical microparticles embosphere 100-300 micrometers (Biosphere Medical, Roissy, France) of the affected joint(s), until partial vascular stasis and decharacterization of pathological synovial enhancement.

These evaluations will be performed at baseline, 1, 3, 6, 12, 24, 36, 48 and 60 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hereditary coagulopathies with arthropathy (i.e., chronic synovitis due to hemarthrosis), with X-ray and MRI (documenting synovitis) followed up at the Hemophilia Center HC-FMUSP.

Exclusion Criteria:

* Patients who do not complete the planned assessments
* Patients who do not accept to continue with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-16 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of synovium thickness by embolization | 6 months
  Measure (in milimeters) changes of synovial thickness in patients with hereditary coagulopathies with arthropathy due to hemarthrosis with MRI (measure synovium thickness)

SECONDARY OUTCOMES:
Reduction of synovitis by embolization | 1, 3 12, 24, 36, 48 and 60 months
  Measure (in milimeters) changes on synovial thickness in patients with hereditary coagulopathies with arthropathy due to hemarthrosis with MRI
Inferior limb strength | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure changes in muscle strength by timed up and go (by time of performance, in seconds).
Inferior limb strength | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure changes in muscle strength of lower limbs by 30 seconds sit to stand test (by number of repetitions)
Balance and fall risk | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure (in seconds, period of time to perform the test) changes in balance and risk of falls by Timed up and go test.
Quality of life of the patient | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure, according to the scale of the questionnaire, changes in quality of life with Haemophilia - Adult - Quality of life Questionnaires (HAEM-A-QoL, 10 dimensions, 0 to 100, being 0 the best health related quality of life)
Quality of life of the patient | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure, according to the scale of the questionnaire, changes in quality of life with Knee Injury and Osteoarthritis Outcome Score (KOOS, 0-100, 100 being the best quality of life).
Quality of life of the patient | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure, according to the scale of the questionnaire, changes in quality of life with by EQ-5D, up to 1, being 1 the best quality of life). Please note: "Since 2009, EQ-5D has been available in three versions: the three-level EQ-5D-3L; the five-level EQ-5D-5L; and a 'youth' adaptation, EQ-5D-Y. Although the EQ is in recognition of the EuroQol group name, the D refers to dimensions, the L signifies level, and the Y stands for youth, the name of the instrument should not be spelled out in this manner as this is inaccurate. Therefore, EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument in general." Brooks R, Boye KS, Slaap B. EQ-5D: a plea for accurate nomenclature. J Patient Rep Outcomes. 2020 Jul 3;4(1):52. doi: 10.1186/s41687-020-00222-9. PMID: 32620995; PMCID: PMC7334333.
Functional capacity | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure (according to the scale of the questionnaire) changes in functional capacity with Functional Independence Score in Hemophilia (FISH score, 0 to 32, 32 being the best result)
Functional capacity | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure (according to the scale of the questionnaire) changes in functional capacity with Functional Independence Score by Knee Injury and Osteoarthritis Outcome Score (KOOS, 0-100, 100 being the best result)
Physical capacity | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure changes in physical capacity by Hemophilia Joint Health Score (HJHS), 0 to 124, 0 being the best result.
Pain of the affected joint | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure changes in pain by Hemophilia Joint Health Score (HJHS, 0-12, 0 being the best result)
Pain of the affected joint | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure changes in pain by numerical rating scale (NRS, 0-10, 0 being no pain and 10 being the worst pain possible)
Pain of the affected joint | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure changes in pain by Knee Injury and Osteoarthritis Outcome Score (KOOS, 0 to 100, 100 being the best result)
Stifness | 1, 3, 6, 12, 24, 36, 48, 60 months
  Measure (0 to 100, 100 being the best result) changes in knee stiffness by Knee Injury and Osteoarthritis Outcome Score (KOOS)

CONTACTS AND LOCATIONS:
Overall Officials: Fabiane E FArias, PT, Principal Investigator — IOT-HC-FMUSP (Orthopedics Institute - General Hospital- School of Medicine - University of Sao Paulo; Andre M Assis, MD, PhD, Study Director — Radiology Insititute, General Hospital, School Medicine, University of São Paulo; Paula Villaça, MD, PhD, Study Director — Hematology department, General Hospital, School of Medicine, University of Sâo Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No